CLINICAL TRIAL: NCT01554189
Title: A Multiple Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of MK-8325 in Hepatitis C Infected Males
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of MK-8325 in Hepatitis C-Infected Males (MK-8325-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8325-002; 2011-006263-22 (EudraCT Number)
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — MK-8325

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Panel A (GT1 10 mg) (Experimental)
  Interventions: Drug: MK-8325
- Panel B (GT1 50 mg) (Experimental)
  Interventions: Drug: MK-8325
- Panel C (GT1 100 mg) (Experimental)
  Interventions: Drug: MK-8325
- Panel D (GT1 200 mg) (Experimental)
  Interventions: Drug: MK-8325
- Panel E (GT3 10 mg) (Experimental)
  Interventions: Drug: MK-8325
- Panel F (GT3 50 mg) (Experimental)
  Interventions: Drug: MK-8325
- Panel G (GT3 100 mg) (Experimental)
  Interventions: Drug: MK-8325
- Panel H (GT3 200 mg) (Experimental)
  Interventions: Drug: MK-8325
- Panel I (GT1a 10 mg) (Experimental)
  Interventions: Drug: MK-8325
- Panel J (GT1a 50 mg) (Experimental)
  Interventions: Drug: MK-8325
- Placebo Panel (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8325 — MK-8325 capsules, orally, once per day for 5 days, at a dose determined by panel assignment (10-200 mg)
  Arms: Panel A (GT1 10 mg); Panel B (GT1 50 mg); Panel C (GT1 100 mg); Panel D (GT1 200 mg); Panel E (GT3 10 mg); Panel F (GT3 50 mg); Panel G (GT3 100 mg); Panel H (GT3 200 mg); Panel I (GT1a 10 mg); Panel J (GT1a 50 mg)
Drug: Placebo — Placebo to match MK-8325 capsules, orally, once per day for 5 days
  Arms: Placebo Panel

SUMMARY:
This study is being done to assess the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of MK-8325 in male hepatitis C virus (HCV)-infected participants. There will be 3 parts to this study. Part I will enroll only genotype 1 (GT1) HCV patients, Part II will enroll only genotype 3 (GT3) HCV-infected participants, and Part III will enroll only GT1a HCV-infected participants. All parts may run concurrently, or may be staggered as needed by the clinical sites.

ELIGIBILITY:
Inclusion criteria:

* Body mass index (BMI) of 18 to ≤37 kg/m^2
* Diagnosis of chronic HCV infection
* Must be infected with HCV GT1a, GT1b, or GT3

Exclusion criteria:

* Co-infection with GT1 and GT3 HCV
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal (excepting HCV infection), cardiovascular, hematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of neoplastic disease
* Positive Hepatitis B surface antigen
* History of human immunodeficiency virus (HIV) infection or positive HIV serology
* Major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior
* History of significant multiple and/or severe allergies (including latex allergy), or anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Current regular user (including "recreational use") of any illicit drugs or history of drug (including alcohol) abuse within approximately 2 months
* Evidence or history of chronic hepatitis not caused by HCV including but not limited to non-HCV viral hepatitis, non-alcoholic steatohepatitis (NASH), drug-induced hepatitis, autoimmune hepatitis
* Previous treatments(s) with nonstructural 5A (NS5A) protein inhibitors
* Treatment with protease inhibitor(s) <30 days prior to study enrollment
* Previous exposure to interferon-alpha and/or ribavirin within 3 months prior to the first dose of MK-8325 in the study
* Clinical or laboratory evidence of advanced or decompensated liver disease; evidence of bridging fibrosis or higher grade fibrosis (Metavir score ≥3) from prior liver biopsy

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 5 in plasma HCV ribonucleic acid (RNA) in GT1 participants | Day 1 predose and 2, 4, 8, 12, 24 and 36 hours post-dose, Days 3 and 4 predose, Day 5 predose and 2, 4, 8, 12, and 24 hours post-dose.
Mean maximum reduction from baseline through Day 5 in HCV ribonucleic acid (RNA) in GT3 participants | Day 1 predose and 2, 4, 8, 12, 24 and 36 hours post-dose, Days 3 and 4 predose, Day 5 predose and 2, 4, 8, 12, and 24 hours post-dose.
Number of participants experiencing at least one adverse event | Day 1 up to 56 days
Number of participants discontinuing study drug due to an adverse event | Days 1-5

SECONDARY OUTCOMES:
Trough plasma concentration (C24hr) of MK-8325 | Day 1 predose and 0.25 0.5, 1, 2, 4, 5, 6, 7, 8, 12, 16 and 24 hours post-dose and Day 5 predose and 0.25, 0.5, 1, 2, 4, 5, 6, 7, 8, 12, 16, 24, 36,48, 72, 96, 120, 144, 168, 192, 216, and 240 hours post-dose
Area under the concentration curve from Hour 0 to Hour 24 (AUC0-24hr) for MK-8325 | Day 1 predose and 0.25 0.5, 1, 2, 4, 5, 6, 7, 8, 12, 16 and 24 hours post-dose and Day 5 predose and 0.25, 0.5, 1, 2, 4, 5, 6, 7, 8, 12, 16 and 24 hours post-dose
Maximum plasma concentration (Cmax) of MK-8325 | Day 1 predose and 0.25 0.5, 1, 2, 4, 5, 6, 7, 8, 12, 16 and 24 hours post-dose and Day 5 predose and 0.25, 0.5, 1, 2, 4, 5, 6, 7, 8, 12, 16, 24, 36,48, 72, 96, 120, 144, 168, 192, 216, and 240 hours post-dose